CLINICAL TRIAL: NCT06065163
Title: Ultrasound Guided Diuretic Therapy in Type 1 Cardiorenal Syndrome
Acronym: NEEDED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Collaborators: EchoNous Inc. (Industry)
Responsible Party: Principal Investigator, Salvador Lopez Gil, Chief of Hemodialysis Unit, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 22-1339
Record Dates: First submitted 2023-09-27; First posted 2023-10-03 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Cardiorenal Syndrome Type 1

STUDY DESIGN:
Intervention Model Description: Experimental, randomized, double-blind, and prospective study
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound Guided Treatment (Experimental): Patients allocated to this will be guided (diuretic treatment) by ultrasound (VExUS) findings
  Interventions: Other: Diuretic de/escalation based on ultrasound findings (VExUS Score)
- Clinical Guided Treatment (Active Comparator): Patients allocated to this will be guided (diuretic treatment) by clinical congestion score (CCS) findings
  Interventions: Other: Diuretic de/escalation based on clinical findings (CCS Score)

INTERVENTIONS:
Other: Diuretic de/escalation based on ultrasound findings (VExUS Score) — Patients allocated in the experimental arm will have diuretic dosing adjusted based on ultrasound findings (VExUS Score)
  Arms: Ultrasound Guided Treatment
Other: Diuretic de/escalation based on clinical findings (CCS Score) — Patients allocated in the experimental arm will have diuretic dosing adjusted based on clinical findings (CCS Score)
  Arms: Clinical Guided Treatment

SUMMARY:
A double-blind, randomized, controlled trial was conducted with the main objective of evaluating if patients with clinical assessment and VExUS reach decongestion faster within a maximum period of 7 days during the hospital stay. Likewise, the study will describe those patients who experience a decrease in serum creatinine (CrS), NT-proBNP at discharge, greater diuretic adjustment, rate of intrahospital readmission, and 30-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Type 1 cardiorenal syndrome in emergency room at Instituto Nacional de Cardiologia Ignacio Chávez

Exclusion Criteria:

* Patients who denied to participate
* Liver disease (cirrohsis)
* Complex congenital heart disease
* Kidney transplant
* Heart transplant
* Severe valvular disease
* Chronic kidney disease KDIGO G5 and G5d
* INTERMACS Score 2

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Decongestion within 7 days | 7 days
  Assess if the ultrasound guided arm achieves faster decongestion

SECONDARY OUTCOMES:
Acutely decompensated heart failure readmission rate | 7 days
  Assess which strategy achieves less readmission rate
Length of hospital stay | 7 days
  Assess which strategy achieves fewer days of hospital stay
Total diuretic dose within 7 days | 7 days
  Assess which strategy has greater diuretic adjustment
Number of participants that initiate kidney replacement therapy | 30 days
  Assess which strategy is associated with kidney replacement therapy
Intrahospital mortality | 30 days
  Assess which strategy achieves less intrahospital mortality
Days alive out of hospital | 1 month
  Assess which strategy achieves more days alive out of hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Cardiología Ignacio Chávez, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Will share the clinical study report and results when they´re available
Supporting Information: CSR
Time Frame: 2 months before finishing the study
Access Criteria: Via email to principal investigator